CLINICAL TRIAL: NCT05885711
Title: Dutch Title: Zelfmanagement Pessarium Project
Brief Title: Self-management Pessary Project
Acronym: ZPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: Z2022098
Record Dates: First submitted 2023-05-11; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; pessary; self-management
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Self-Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self-management — self-managing a pessary: removing, cleaning and inserting

SUMMARY:
The goal of this multicenter observational study is to study self-management of pessary therapy in patients with pelvic organ prolapse.

The primary question it aims to answer is:

• how many patients succeed learning self-management if offered a standardized training?

Secondary outcomes are:

* how many patients are willing to learn self-management?
* what patient factors contribute to successfully learning self-management and willingness to self-manage?
* how satisfied are patients with pessary therapy and self-management?
* the occurrence of side-effects
* continuation and quitting of pessary therapy and self-management
* cross-over to surgery
* number of visits to doctor because of pessary therapy
* healthcare costs

Participants will be asked to fill in questionnaires three times during the study (upon inclusion, 6 weeks and 12 months after starting self-management or after starting pessary therapy with a correctly fitting pessary).

Researchers will compare the self-managing patient to the non-self-managing patients.

ELIGIBILITY:
Inclusion Criteria:

* fitted a ring, sieve of knob pessary
* above 18 years old
* able to understand patient information

Exclusion Criteria:

* fitted a new pessary to replace an old one (continuing former pessary therapy)
* fitted a new pessary after they experienced adverse effects of a former pessary

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: New patients that get fitted a pessary in second line (hospital)
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that succeed in learning self-management of the pessary | immediately after self-management training, it is determined whether patients can remove and insert their pessary
  Patients were offered self-management training, after explanation they were asked to remove and insert their pessary twice. Succes was defined as removing and inserting the pessary completely independent the second time.

CONTACTS AND LOCATIONS:
Overall Officials: M Weemhoff, Principal Investigator — Zuyderland Medisch Centrum
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided